CLINICAL TRIAL: NCT06230926
Title: Turkish Adaptation, Validity and Reliability of "Parkinson's Disease Quality of Life 7 (PDQoL7)" Questionnaire
Brief Title: Turkish Adaptation of "Parkinson's Disease Quality of Life 7 (PDQoL7)" Questionnaire
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Asli Demirtaş, Lecturer, PT. MSc., Nigde Omer Halisdemir University
Other Study IDs: Gazi University-05.09.2023.2
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease; Quality of Life
Keywords: Parkinson's disease; Qality of life; Patient Reported Measure; Validity; Reliability; Adaptation
MeSH Terms: conditions — Parkinson Disease | interventions — Acclimatization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease Group: The study will be conducted in collaboration with Gazi University Faculty of Health Sciences and Niğde Ömer Halisdemir University. The study data will be obtained from individuals diagnosed with PD admitted to the Neurology Outpatient Clinic of Niğde Ömer Halisdemir University Training and Research Hospital. Necessary permissions were obtained from all institutions and questionnaire developers. Since at least 5-10 times the number of items in the questionnaire (7 items) must include at least 5-10 times the number of participants in order to perform factor analysis, a pretest of the questionnaire will be applied to individuals with PD with at least 35-70 participants.
  Interventions: Other: Validity, Reliability and Adaptation

INTERVENTIONS:
Other: Validity, Reliability and Adaptation — The Hoehn & Yahr Scale (HDS) and the Unified Parkinson's Disease Rating Scale (UPDRS) will be used for the clinical evaluation and disease staging of the individuals included in the study. In addition to the PDQoL-7 questionnaire, the 'Short Form-36' and 'Parkinson's Disease Questionnaire-39' questionnaires will be administered to patients to assess concurrent validity. Since at least 5-10 times the number of items in the questionnaire (7 items) must include at least 5-10 times the number of participants in order to perform factor analysis, a pretest of the questionnaire will be applied to individuals with PD with at least 35-70 participants. To determine the test-retest reliability, the PDQoL7 questionnaire will be administered again to the same patients after 2 weeks.

SUMMARY:
Parkinson's Disease (PD) is a progressive neurodegenerative disorder characterized by the involvement of dopaminergic pathways in the basal ganglia. Motor and non-motor symptoms are frequently observed in PD. These symptoms may negatively affect the quality of life of individuals with PD. Therefore, it is recommended to evaluate the quality of life of individuals with PD and plan appropriate treatments. The "Parkinson's Disease Quality of Life 7 (PDQoL7)" questionnaire is a patient-reported quality of life assessment questionnaire developed specifically for individuals with PD. The questionnaire, which consists of 7 questions in total, evaluates the degree of difficulty the patient has in performing various activities. The aim of this study was to adapt the PDQoL7 questionnaire into Turkish and to establish its validity and reliability.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a progressive neurodegenerative disorder characterized by the involvement of dopaminergic pathways in the basal ganglia. Motor and non-motor symptoms are frequently observed in PD. These symptoms may negatively affect the quality of life of individuals with PD. Therefore, it is recommended to evaluate the quality of life of individuals with PD and plan appropriate treatments. The "Parkinson's Disease Quality of Life 7 (PDQoL7)" questionnaire is a patient-reported quality of life assessment questionnaire developed specifically for individuals with PD. The questionnaire, which consists of 7 questions in total, evaluates the degree of difficulty the patient has in performing various activities. The aim of this study was to adapt the PDQoL7 questionnaire into Turkish and to establish its validity and reliability. The study data will be collected in collaboration with Gazi University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation and Niğde Ömer Halisdemir University and will be conducted with individuals diagnosed with PD who applied to the Neurology Outpatient Clinic of Niğde Ömer Halisdemir University Training and Research Hospital. Necessary permissions were obtained from all institutions and the people who developed the questionnaire. After the purpose and method of the study were explained to the participants in detail, individuals who voluntarily agreed to participate in the study will be included in the study. The serial approach method will be used when translating the original questionnaire into Turkish. Since at least 5-10 times the number of items in the questionnaire should be included in order to perform factor analysis, a pretest of the questionnaire will be applied to individuals with PD with at least 35-70 participants. "Parkinson's Disease Questionnaire-39" and "Short Form-36" questionnaires will be administered to the patients to assess concurrent validity. To determine test-retest reliability, the PDQoL7 questionnaire will be administered to the same patients 2 weeks later, and correlation analysis and test-retest reliability will be calculated. Cronbach's Alpha Reliability coefficient will be applied to determine the internal consistency of the questionnaire. The construct validity of PDQoL7 will be analyzed by confirmatory factor analysis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with PD by a neurologist,
* Understands and speaks Turkish,
* Individuals who score 18 points or above from the mini-mental state assessment will be included.

Exclusion Criteria:

* People with dementia, hearing and/or vision loss
* Patients who are illiterate will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research will be carried out in cooperation with Gazi University Faculty of Health Sciences and Niğde Ömer Halisdemir University. Study data will be obtained from individuals diagnosed with PD who apply to Niğde Ömer Halisdemir University Training and Research Hospital Neurology Polyclinic. Necessary permissions were obtained from all institutions and those who developed the survey.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Quality of Life 7 Questionnaire (PDQoL7) | Baseline
  The questionnaire assesses the quality of life of individuals with PD in the last week based on patient self-report. The questionnaire consists of a total of 7 questions and is answered on a 5-point Likert scale ranging from 0 (never)-4 (always). The total score varies between 0 and 28 points and the higher the score, the more negatively the patients' quality of life is affected.
Parkinson's Disease Questionnaire-39 (PDQ-39) | Baseline
  The Parkinson's Disease Questionnaire (PDQ-39) is the most commonly used questionnaire to assess health-related quality of life specific to PD. The PDQ- 39 includes 39 questions in 8 different domains; mobility (10 questions); activities of daily living (6 questions); emotional state (6 questions); stigma (4 questions); social support (3 questions); cognition (4 questions); communication (3 questions); and physical pain (3 questions). Questions are answered with the last 1 month in mind. For each question, a score is given from 0: no problem at all to 4: constant problem. The lower the total score, the better the quality of life. It is a quality of life questionnaire developed specifically for Parkinson's disease.
Short-Form 36 (SF-36) | Baseline
  SF-36 evaluates the negative and positive aspects of health status. The 8 subscales of the scale consist of a total of 36 questions including I-physical function (10 items), II-social function (2 items), III- role limitation due to physical problems (4 items), IV- role limitation due to emotional problems (3 items), V- mental status (5 items), VI- energy/vitality (4 items), VII-pain (2 items), VIII- general perception of health (5 items). The scores of the subscales range from 0 to 100 (0: indicating poor health status, 100: indicating no problem in health status). As a result, it is possible to obtain separate scores for each subscale. The answers to the items are asked to be based on the person's condition in the last 4 weeks.

SECONDARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline
  MMSE will be used to evaluate cognitive functions. The mini mental test is categorized under five main headings. It consists of 11 items including orientation (10 points), recording memory (3 points), attention and calculation (5 points), recall (3 points) and language (9 points). It is evaluated over 30 points in total. A score between 24-30 points is defined as normal, 18-23 points as mild dementia, and 17 points and below as severe dementia. The average administration time of the test is 10 minutes. Patients scoring 18 and above will be included in the study.
Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline
  Unified Parkinson's Disease Rating Scale (UPDRS) is a scale created to evaluate the motor performance, mental and spiritual status, and daily life activities of patients diagnosed with PD. The scale consists of a total of 4 sections and 42 items. In the first part, non-motor symptoms such as thoughts, behavior and affect; In the second part, activities of daily living; motor symptoms in the third part; In the fourth section, treatment complications are evaluated. Each item is scored between 0 (no symptoms or signs) and 4 (the most severe symptom or sign possible).
Modified Hoehn-Yahr Evaluation (MHYE) | Baseline
  Modified Hoehn-Yahr Evaluation (MHYE) used to define the disease stage of patients diagnosed with PD. According to MHYE, the disease consists of 8 stages. It is stated that the disease symptoms worsen as the stage progresses.
Interview Form | Baseline
  All evaluations will be carried out by face-to-face interview method. Individual characteristics of the patients (gender, age, height, body weight, marital status, education level, dominant extremity, smoking and alcohol consumption habits, use and type of assistive device, how many years the assistive device has been used) and disease-related (year of diagnosis, disease duration Information (such as CV, family history, medications used, surgeries) will be questioned.

CONTACTS AND LOCATIONS:
Overall Officials: İlke KESER, Prof. Dr., Study Director — Gazi University
Locations (3):
- Turkey (Türkiye) (3):
  - Ankara Medipol University, Ankara
  - Gazi University, Ankara
  - Niğde Ömer Halisdemir University, Niğde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stathis P, Papadopoulos G. Evaluation and validation of a patient-reported quality-of-life questionnaire for Parkinson's disease. J Patient Rep Outcomes. 2022 Mar 2;6(1):17. doi: 10.1186/s41687-022-00427-0. PMID 35235090
- [Background] Zhao N, Yang Y, Zhang L, Zhang Q, Balbuena L, Ungvari GS, Zang YF, Xiang YT. Quality of life in Parkinson's disease: A systematic review and meta-analysis of comparative studies. CNS Neurosci Ther. 2021 Mar;27(3):270-279. doi: 10.1111/cns.13549. Epub 2020 Dec 28. PMID 33372386
- [Background] Fereshtehnejad SM. Strategies to maintain quality of life among people with Parkinson's disease: what works? Neurodegener Dis Manag. 2016 Oct;6(5):399-415. doi: 10.2217/nmt-2016-0020. Epub 2016 Sep 7. PMID 27600287